CLINICAL TRIAL: NCT01237769
Title: Effect of Vitamin D on Metabolic Parameters in Patients With the Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Prof Moses Elisaf, University of Ioannina Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2010-11

CONDITIONS: Metabolic Syndrome
Keywords: vitamin D; Metabolic syndrome; Hypertension; Dyslipidemia; Dysglycemia; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Dyslipidemias; Inflammation | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): All patients will be instructed to exercise and lose weight according to the NCEP-ATP III diet. The participants will be randomized in an open manner into one of the following 2 treatment groups: a) cholecalciferol (VitD3) (2200 IU/day) plus lifestyle measures or b) only lifestyle measures. Recruitment will be completed within one year. The reassessment of the patients will be done 3 months after starting of treatment.
  Interventions: Drug: Vitamin D3
- Lifestyle measures (Active Comparator)
  Interventions: Behavioral: Lifestyle advice

INTERVENTIONS:
Drug: Vitamin D3 — 2200 IU/day
  Other Names: vitamin D
  Arms: Vitamin D
Behavioral: Lifestyle advice — Diet and exercise
  Other Names: Lifestyle measures
  Arms: Lifestyle measures

SUMMARY:
In recent years emphasis has been given to investigate the role of vitamin D in areas beyond bone metabolism and maintenance of calcium homeostasis. Thus, vitamin D deficiency has been associated with risk factors for the occurrence of cardiovascular disease as well as with overall mortality.In addition, there are indications that a large proportion of the population (up to 50%) is vitamin D deficient. The measurement of vitamin 25 (OH) D3 levels is the best way to estimate the vitamin D actual reserves. It is worth mentioning that elevated levels of parathyroid hormone (PTH) [5] and reduced levels of 1,25 (OH)2 vitamin D3 (calcitriol have also been associated with cardiovascular disease.

The metabolic syndrome is a sum of risk factors for cardiovascular disease and is found in approximately 25% of the Greek population.There are a lot of data linking low vitamin D levels with the metabolic syndrome as a whole as well as with its individual characteristics. Specifically, vitamin D deficiency has been associated with increased incidence of hypertension, dyslipidemia, obesity, inflammation and dysglycemia.

Many studies have explored the effect of giving vitamin D supplements on the risk factors associated with the metabolic syndrome and the cardiovascular disease. The results of these studies are conflicting and this may partially be due to different doses of vitamin D used. The form of vitamin D most commonly used in these studies is cholecalciferol (vitamin D3.

Aim of the study:

Determination of the effect of cholecalciferol (VitD3) (2200 IU/day) on metabolic parameters in patients with metabolic syndrome.

Endpoints:

The primary endpoint will be changes in metabolic syndrome parameters 3 months after starting treatment:

* Waist circumference
* Blood pressure
* Levels of fasting serum triglycerides
* Levels of high-density lipoprotein cholesterol (HDL-C)
* Levels of fasting serum glucose.

The secondary endpoints will include changes in:

* The levels of low-density lipoprotein cholesterol (LDL-C) and non-HDL-C
* Subfractions of LDL-C [average particle size of LDL-C, levels of small dense (sd) LDL-C]
* Subfractions of HDL-C (levels of small and large particle HDL-C)
* The activity and levels of Lp-PLA2 (lipoprotein-associated phospholipase A2)
* The levels of serum apolipoprotein AI, A-II, AV, B, E, C-II, C-III and lipoprotein (Lp) (a)
* The activity of paraoxonase-1 (PON1)
* The concentration of pre-beta1-HDL
* The levels of hs-CRP (high sensitivity C-reactive protein)
* Oxidative stress as measured by levels of 8-isoprostane in the blood and urine and oxidized LDL (oxLDL)
* Adipokine levels (leptin, adiponectin, visfatin)
* Glucose homeostasis (index HOMA: fasting insulin X fasting glucose/405)
* The levels of glycosylated hemoglobin (HbA1c)
* The levels of 25 (OH) vitamin D3, of 1,25 (OH)2 vitamin D3 and PTH
* The levels of serum electrolytes (Ca, PO4) and the activity of alkaline phosphatase (ALP) in serum.

Study population:

The investigators will study patients with metabolic syndrome (n = 50 adults) attending the Outpatient Lipid and Obesity clinic at the University Hospital of Ioannina. Diagnosis of the Metabolic Syndrome will be based on the criteria of National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATP III).

All patients will be instructed to exercise and lose weight according to the NCEP-ATP III diet. The participants will be randomized in an open manner into one of the following 2 treatment groups: a) cholecalciferol (VitD3) (2200 IU/day) plus lifestyle measures or b) only lifestyle measures. Recruitment will be completed within one year. The reassessment of the patients will be done 3 months after starting of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metabolic syndrome (n = 50 adults) attending the Outpatient Lipid and Obesity clinic at the University Hospital of Ioannina. Diagnosis of the Metabolic Syndrome will be based on the criteria of National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATP III).

Exclusion Criteria:

* The study will exclude patients with triglyceride levels >500 mg/dL,
* Diabetes mellitus, hypothyroidism (TSH >5 IU/mL),
* Primary hyperparathyroidism, hypercalcemia of any cause,
* A history of taking formulations of calcium or vitamin D,
* Alcohol consumption >3 drinks per day for men and >2 drinks per day for women and women of childbearing age not taking contraceptive measures.
* Patients with hypertension may be included in the study if their blood pressure is <140/90 and the antihypertensive treatment remains constant over the past 3 months (no change of antihypertensive medication during the study).
* Finally, patients receiving lipid-lowering medicines or patients who have stopped taking them for less than 4 weeks will be excluded from the study.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic syndrome incidence 3 months after starting treatment | Baseline and 3 months

SECONDARY OUTCOMES:
Change in levels of fasting glucose | Baseline and 3 months
Change in levels of high-density lipoprotein cholesterol (HDL-C) | Baseline and 3 months
Change in levels of blood pressure | Baseline and 3 months
Changes in serum triglycerides | Baseline and 3 months
Changes in levels of low-density lipoprotein cholesterol (LDL-C) | Baseline and 3 months
Changes in levels of small dense low-density lipoprotein cholesterol (sdLDL-C) | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Moses Elisaf, MD, Principal Investigator — University of Ioannina Medical School
Locations (1):
- Outpatient Lipid Clinic, University Hospital of Ioannina, Ioannina, Ioannina, Greece

REFERENCES:
- [Derived] Makariou SE, Elisaf M, Challa A, Tellis C, Tselepis AD, Liberopoulos EN. Effect of combined vitamin D administration plus dietary intervention on oxidative stress markers in patients with metabolic syndrome: A pilot randomized study. Clin Nutr ESPEN. 2019 Feb;29:198-202. doi: 10.1016/j.clnesp.2018.10.004. Epub 2018 Oct 24. PMID 30661687
- [Derived] Makariou SE, Elisaf M, Challa A, Tentolouris N, Liberopoulos EN. No effect of vitamin D supplementation on cardiovascular risk factors in subjects with metabolic syndrome: a pilot randomised study. Arch Med Sci Atheroscler Dis. 2017 Oct 5;2:e52-e60. doi: 10.5114/amsad.2017.70504. eCollection 2017. PMID 29242845
- See also: Related Info — http://www.bpath.gr